CLINICAL TRIAL: NCT04378010
Title: A Phase 2b Randomized, Double-Blind, Placebo-controlled, Multicenter Study Evaluating Safety and Efficacy of EDP-305 in Subjects With Liver Biopsy Proven Non-alcoholic Steatohepatitis (NASH) (ARGON-2)
Brief Title: A Randomized, Double-blind Study to Assess the Safety and Efficacy of EDP-305 in Subjects With Liver-biopsy Proven NASH
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Enanta Pharmaceuticals, Inc. made the strategic decision to discontinue the ARGON-2 study to prioritize combination treatment approaches. This decision was not based on safety concerns.
Sponsor: Enanta Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EDP 305-102; 2019-003876-38 (EudraCT Number)
Record Dates: First submitted 2020-05-04; First posted 2020-05-07 (Actual); Results first posted 2023-05-19 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-04

CONDITIONS: Non-Alcoholic Steatohepatitis
Keywords: Fatty Liver, non-alcoholic fatty liver disease, NASH
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fatty Liver | interventions — EDP-305

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- EDP-305 1.5 mg (Experimental): Once a day orally for 72 weeks
  Interventions: Drug: EDP-305 1.5 mg
- EDP-305 2 mg (Experimental): Once a day orally for 72 weeks
  Interventions: Drug: EDP-305 2 mg
- Placebo (Placebo Comparator): Once a day orally for 72 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: EDP-305 1.5 mg — Tablet
  Other Names: EDP-305
  Arms: EDP-305 1.5 mg
Drug: EDP-305 2 mg — Tablet
  Other Names: EDP-305
  Arms: EDP-305 2 mg
Drug: Placebo — Tablet
  Arms: Placebo

SUMMARY:
A randomized, double-blind study to assess the safety and efficacy of EDP-305 in subjects with liver-biopsy proven Non-Alcoholic Steatohepatitis (NASH)

DETAILED DESCRIPTION:
The aim of this Phase 2b study aimed to evaluate safety and efficacy of the investigational novel FXR agonist, EDP-305, in a population of patients with liver biopsy proven NASH.

This Phase 2b study aimed to evaluate the safety and efficacy of two doses of EDP-305 compared to placebo for the treatment of NASH in subjects with liver biopsy proven NASH. As suggested in the FDA guidance, this late stage Phase 2 study explored the effect of EDP-305/placebo treatment on histological endpoints. The patient population selected for inclusion in the study was designed to represent the target population for treatment. Specifically, in patients with liver disease, there is a significant overlap of NASH and various metabolic conditions including obesity and T2DM. In order to be reflective of the NASH population, these patients were not excluded from participation in this study.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent documentation signed and dated by the participant.
* Male and female participants, of all ethnic origins, between the ages of 18 and 75 years, inclusive.
* Participants of all ethnic origins had to have a Body Mass Index (BMI) > 25 kg/m2 and ≤ 45 except Asian participants who qualified for the study with BMI > 23 kg/m2.
* Histological evidence of definite NASH based on NASH Clinical Research Network (CRN) criteria obtained from assessment of a liver biopsy by the central histopathologist. The biopsy may be obtained either 1) during the Screening window or 2) within 26 weeks prior to the Screening visit.
* NAFLD Activity Score (NAS) of 4 or greater with a score of at least 1 in each component of the NAS (steatosis scored 0-3, lobular inflammation scored 0-3, ballooning scored 0-2).
* Fibrosis stage 2 or 3 using the NASH CRN Histologic Scoring System.
* Participants had to have Screening laboratory values for Hepatitis B surface antigen (HBsAg), anti-HCV antibodies and HCV RNA, and Human Immunodeficiency Virus (HIV) 1 and 2 antibodies (Ab) as seronegative. [Note: participants previously infected by chronic hepatitis C and treated with direct acting antivirals (DAAs) with sustained virologic response (SVR) for at least 3 years were allowed.]
* A woman of childbearing potential who was sexually active with a male had to agree to use two effective methods of contraception from the date of Screening until 30 days after the last dose of study drug.
* A male participant who had not had a vasectomy and was sexually active with a woman of childbearing potential had to agree to use effective contraception from the date of Screening to 90 days after the last dose of study drug.
* Participant had to be willing and able to adhere to the assessments, visit schedules, prohibitions and restrictions, as described in this protocol.

Exclusion Criteria:

* Laboratory Screening results as indicated below:

  * Total white blood cells (WBC) <3000 cells/mm3
  * Absolute neutrophil count (ANC) <1500 cells/mm3
  * Platelet count <140,000/mm3
  * International Normalized Ratio, INR >1.2 (unless due to use of anticoagulants)
  * Estimated glomerular filtration rate (eGFR) < 60 mL/min according to the Modification of Diet in Renal Disease (MDRD) equation
  * AST ≥5× ULN
  * ALT ≥5× ULN
  * ALP ≥2× ULN
  * Total bilirubin > 1.5 times ULN during Screening. [Note: Patients with Gilbert's syndrome were allowed following review by the Medical Monitor if they had a known history of Gilbert's syndrome with a normal direct bilirubin value and normal reticulocyte count.]
* Pregnant or nursing females.
* MELD: Model for End-stage Liver Disease score >12.
* Clinical or laboratory evidence of known chronic liver disease such as alcoholic liver disease, primary biliary cholangitis (PBC), primary sclerosing cholangitis (PSC), autoimmune hepatitis, Wilson disease, iron overload, alpha-1-antitrypsin deficiency, drug-induced liver injury, known or suspected hepatocellular carcinoma (HCC).
* History of acute liver complications due to gallstones (e.g., acute cholecystitis or acute biliary obstruction) unless the participant had a cholecytectomy (more than 3 months prior to screening).
* History of liver transplant, or current placement on a liver transplant list.
* Hepatorenal syndrome (type I or II).
* Prior variceal hemorrhage, uncontrolled encephalopathy, liver cirrhosis Child-Pugh Class A, B, and C, esophageal varices, or refractory ascites within the previous 26 weeks of Screening and/or histological presence of liver cirrhosis.
* Prior or planned ileal resection, or prior or planned bariatric surgery. [Note: Participants who had undergone gastric surgeries that did not affect drug absorption (e.g., gastric band or gastric sleeve procedures) were allowed if they were stable for at least 1 year prior to Screening. Gastrectomy or Roux-en-Y bypass was allowed if stable for at least 3 years prior to Screening.]
* Participants with clinically or otherwise documented cardiovascular or cerebrovascular disease including clinically significant anomalies of rhythm or pattern of ECG, that in the judgement of the Principal Investigator (PI) could affect the safety of the participant or their ability to comply with the study requirements.
* HbA1c ≥ 9.5% within 60 days prior to Day 1.
* Use of a new antidiabetic regimen in the months prior to Screening including metformin, glucagon-like peptide (GLP) 1 agonists, sodium glucose cotransporter-2 (SGLT2) inhibitors, sulfonylureas, or dipeptidyl peptidase 4 (DPP4) inhibitors, insulin or peroxisome proliferator-activated receptor (PPAR)γ agonists (e.g., pioglitazone or rosiglitazone). For pre-existing antidiabetic treatment, participants were to be on a stable dose of antidiabetic drugs: (1) for at least 8 weeks (for metformin and/or sulfonylureas), (2) 12 weeks (for SGLT2 or DPP4 inhibitors), or (3) 12 weeks (for GLP-1 receptor agonists and thiazolidinediones) prior to Screening with the intention to keep the regimen stable during the study.
* Use of a new statin regimen or other lipid lowering agents from 12 weeks prior to Screening.
* Use of a new fibrate regimen from 12 weeks prior to Screening.
* Participants with contraindications to MRI imaging, or not being able to have the MRI performed.
* Participant had received any investigational agent (including investigational vaccine) or biological product within 30 days or 5 times the half-life (whichever was longer) prior to the planned first dose of study drug.
* Use of an experimental or approved treatment for NASH within 26 weeks of Screening.
* Prior use of OCA within 26 weeks of Screening and/or concurrent treatment with OCA (or any other FXR agonists).
* Use of systemic immunosuppressant (e.g., corticosteroids) for more than 4 weeks in duration within 1 year prior to Screening with the intention to continue during the study (chronic use of inhaled, topical, ophthalmological, nasal corticosteroids was allowed)
* Use of any prohibited concomitant medications, including systemic CYP3A4 inhibitors and inducers, within 14 days prior to the first dose of study drug and for the duration of the study.
* Clinically significant history of drug sensitivity or drug allergy, as determined by the PI.
* Current or history of significant alcohol consumption defined as: >14 standard drinks per week and/or ≥4 standard drinks per occasion for males and >7 standard drinks per week and/or ≥3 standard drinks per occasion for females.
* History of substance (including alcohol) abuse and in the judgement of the PI, the participant was not suitable for participation in the study.
* Any other condition(s) that would compromise the safety of the participant or compromise the quality of the clinical study, as judged by the PI.
* Use of medication for weight loss or appetite reduction (e.g., orlistat, bupropion/naltrexone, phentermine-topiramate, phentermine, lorcaserin, non-prescription supplements) at Screening.
* History of malignancy of any organ system (other than localized and considered cured cutaneous basal or squamous cell carcinoma, or in situ cervical cancer), treated or untreated, within 5 years of Screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2020-01-27 (Actual); Primary Completion 2021-10-04 (Actual); Study Completion 2021-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Enanta Pharmaceuticals, Inc, Study Director — Enanta Pharmaceuticals, Inc
Locations (81):
- United States (68):
  - Arizona Liver Health, Chandler, Arizona
  - The Institute of Liver Health, Glendale, Arizona
  - Dignity Health DBA St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Del Sol Research Management LLC, Tucson, Arizona
  - Rajeev Krishan, MD, Inc, Bakersfield, California
  - eStudy Site, Chula Vista, California
  - Southern California Research Center, Coronado, California
  - St. Jude Hospital Yorba Linda DBA St. Joseph Heritage Healthcare, Fullerton, California
  - National Institute of Clinical Research, Inc, Garden Grove, California
  - eStudySite - La Mesa, La Mesa, California
  - Om Research LLC, Lancaster, California
  - Keck Medical Center Of USC, Los Angeles, California
  - Inland Empire Liver Foundation, Rialto, California
  - UC Davis Medical Center, Sacramento, California
  - Southern California Gastrointestinal and Liver Centers, San Clemente, California
  - Precision Research Institute, Llc, San Diego, California
  - Paradigm Clinical Research Institute, Torrance, California
  - Universal Axon Clinical Research, Doral, Florida
  - Fleming Island Center for Clinical Research, Fleming Island, Florida
  - Universal Axon- Homestead, LLC, Homestead, Florida
  - Nature Coast Clinical Research, Inverness, Florida
  - Westside Center for Clinical Research, Jacksonville, Florida
  - Jacksonville Center for Endoscopy - Southside ; Borland Groover Clinic, Jacksonville, Florida
  - Encore Borland Groover Clinical Research, Jacksonville, Florida
  - Meridien Research, Lakeland, Florida
  - Meridien Research, Maitland, Florida
  - Research Associates of South Florida, Miami, Florida
  - University of Miami, Miller School of Medicine-Don Soffer Clinical Research Center, Miami, Florida
  - Well Pharma Medical Research, Corp., Miami, Florida
  - Med Research Of Florida, LLC, Miami, Florida
  - San Marcus Research Clinic, Inc., Miami Lakes, Florida
  - Ocala GI Research, Ocala, Florida
  - IMIC, Inc., Palmetto Bay, Florida
  - Meridien Research, St. Petersburg, Florida
  - Guardian Angel Research, Tampa, Florida
  - Agile Clinical Research Trials, LLC, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center - University Cardiovascular Surgeons, Chicago, Illinois
  - Digestive Research Alliance of Michiana, South Bend, Indiana
  - University Of Iowa Hospital & Clinics, Iowa City, Iowa
  - Ochsner Health System, New Orleans, Louisiana
  - University of Maryland, Baltimore, Maryland
  - Mercy Medical Center, Baltimore, Maryland
  - Digestive Disease Associates, PA, Catonsville, Maryland
  - Mid-Atlantic GI Research, Greenbelt, Maryland
  - Henry Ford Health Hospital, Detroit, Michigan
  - Southern Therapy and Advanced Research LLC GI Associates and Endoscopy Center, Jackson, Mississippi
  - St. Louis Univ. School Of Medicine, St Louis, Missouri
  - AGA Clinical Research Associates, LLC, Egg Harbor, New Jersey
  - Intercity Gastroenterology, Fresh Meadows, New York
  - New York University Medical Centre, New York, New York
  - University of Rochester Medical Center School of Medicine and Dentistry, Rochester, New York
  - Northeast GI Research Division, Concord, North Carolina
  - Carolinas HealthCare System Digestive - Huntersville, Huntersville, North Carolina
  - Lucas Research, Morehead City, North Carolina
  - Cleveland Clinic - Taussig Cancer Institute, Cleveland, Ohio
  - University of Pittsburgh Medical Center - Center for Liver Diseases, Pittsburgh, Pennsylvania
  - Digestive Health Research, LLC, Hermitage, Tennessee
  - Digestive Health Research, Lebanon, Tennessee
  - Quality Medical Research, Nashville, Tennessee
  - Texas Clinical Research Institute, Arlington, Texas
  - Texas Diabetes & Endocrinology, Austin, Texas
  - Crescent Health Clinical, DeSoto, Texas
  - DHAT Research Institute, Garland, Texas
  - American Research Corporation at The Texas Liver Institute, San Antonio, Texas
  - Clinical Trials of Texas, Inc., San Antonio, Texas
  - Bon Secours St. Mary's Hospital of Richmond, Inc, Newport News, Virginia
  - Liver Institute Northwest, Seattle, Washington
- CINME, Buenos Aires, Buenos Aires F.D., Argentina
- University of Calgary, Calgary, Alberta, Canada
- Germany (2):
  - Klinikum der Johann Wolfgang Goethe-Universitaet Frankfurt, Frankfurt am Main, Hesse
  - Universitaetsmedizin der Johannes Gutenberg Universitaet Mainz KoeR, Mainz, Rhineland-Palatinate
- Latin Clinical Trial Center, San Juan, Puerto Rico
- United Kingdom (8):
  - MediNova West London Quality Research Site, Wokingham, Berkshire
  - MeDiNova East London Quality Research Site, Romford, Essex
  - King's College Hospital - King's College Hospital NHS Foundation Trust, London, Greater London
  - MeDiNova South London Quality Research Site, Sidcup, Kent
  - MeDiNova Northampton Dedicated research site, Corby, Northamptonshire
  - MeDiNova Warwickshire Quality Research Site, Kenilworth, Warwickshire
  - MeDiNova Yorkshire Quality Research Site, Shipley, Yorkshire
  - MeDiNova North London Quality Research Site, Middlesex

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Male and female subjects with liver biopsy proven NASH between the ages of 18 and 75 years, inclusive, and with a NAS of 4 or greater with a score of at least 1 in each component of the NAS (steatosis scored 0-3, lobular inflammation scored 0-3, ballooning scored 0-2) and fibrosis stage 2 or 3 using the NASH Clinical Research Network (CRN) Histologic Scoring System were eligible for inclusion. Subjects had to be negative for hepatitis B, hepatitis C, and human immunodeficiency virus (HIV).
Pre-assignment Details: Screening assessments were conducted within 70 days prior to the first dose of study drug (i.e., Study Days -70 to -1). Screening assessments were performed and confirmed sequentially as follows: a) medical history and other noninvasive assessments, b) laboratory assessments, c) MRI-PDFF and MRE and, lastly, d) liver biopsy.
Period: Overall Study
Arm/Group | EDP-305 1.5 mg | EDP-305 2 mg | Placebo
Started | 32 | 34 | 32
Completed | 0 | 0 | 0
Not Completed | 32 | 34 | 32
Not completed — Adverse Event | 8 | 14 | 4
Not completed — Withdrawal by Subject | 0 | 2 | 1
Not completed — Protocol Violation | 2 | 1 | 4
Not completed — Study terminated by Sponsor | 22 | 16 | 22
Not completed — Subject inability to complete study visit | 0 | 0 | 1
Not completed — Subject never dosed | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: NOTE: In the EDP-305 2mg arm 1 participant was randomized but not treated.
Groups:
- Total: Total of all reporting groups
Arm/Group | EDP-305 1.5 mg | EDP-305 2 mg | Placebo | Total
Number analyzed (Participants) | 32 | 33 | 32 | 97
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 22 | 27 | 27 | 76
  >=65 years | 10 | 6 | 5 | 21
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.7 (12.67) | 56.2 (8.14) | 52.7 (11.33) | 56.0 (10.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 19 | 19 | 58
  Male | 12 | 14 | 13 | 39
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 2 | 3 | 2 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 2 | 4
  White | 29 | 27 | 28 | 84
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Argentina | 1 | 0 | 0 | 1
  Canada | 1 | 0 | 0 | 1
  United States | 30 | 31 | 31 | 92
  United Kingdom | 0 | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants Who Achieve ≥1 Stage Improvement in Fibrosis Without Worsening of Steatohepatitis and/or Resolution of Steatohepatitis and no Worsening of Liver Fibrosis as Determined by Liver Biopsy
Description: Proportion of participants who achieve ≥1 stage improvement in fibrosis without worsening of steatohepatitis and/or resolution of steatohepatitis and no worsening of liver fibrosis as determined by liver biopsy.
Time Frame: Week 72
Population: Due to study termination, the biopsy at Week 72 was not performed for any participant. Hence, there were no results to report.
Arm/Group | EDP-305 1.5 mg | EDP-305 2 mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Change in 5D-itch Scale From Baseline
Description: 5D-itch scale, change from baseline at Week 12. Change from baseline for 5D-itch scale was analyzed using a restricted maximum likelihood-based mixed model repeated measures (MMRM) technique. The model included treatment, visit, treatment-by-visit interaction as fixed effects along with baseline NAS score and baseline score for 5D-itch scale as covariate.
  A multidimensional 5D-itch scale developed by Elman (Elman et al., 2010) indicated sum of 0-2 = score of 1, sum of 3-5 = score of 2, sum of 6-10 = score of 3, sum of 11-13 = score of 4, and sum of 14-16 = score of 5. The total 5D score was obtained by summing up the five domain scores and ranges between 5 (no pruritus) and 25 (most severe pruritus).
Time Frame: Baseline, Week 12
Population: ITT population: Intent-to-treat population (ITT) defined as all participants who randomized to treatment. Participants were analyzed according to the treatment to which they were randomized. The overall numbers of participants by group were N = 32, N = 33, and N = 32. The numbers of participants with available data for the specified time frame were n = 7, n = 6 and n = 7 for EDP-305 1.5, 2mg and Placebo groups, respectively, presented as LS Mean (95% CI).
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Placebo: Once a day orally for 72 weeks Placebo: Tablet
Arm/Group | EDP-305 1.5 mg | EDP-305 2 mg | Placebo
Number analyzed (Participants) | 7 | 6 | 7
score on a scale | 2.275 [-1.227 to 5.777] | 4.594 [0.676 to 8.513] | 2.714 [-0.955 to 6.384]
Statistical Analysis 1: Comparison: EDP-305 2 mg vs Placebo; Test type: Other; p = 0.454, Mixed model repeated measures; LS mean difference = 1.880, 95% CI 2-sided [-3.479 to 7.239], Standard Error of Mean 1.788
Statistical Analysis 2: Comparison: EDP-305 1.5 mg vs Placebo; Test type: Other; p = 0.848, Mixed model repeated measures; LS mean difference = -0.439, 95% CI 2-sided [-5.458 to 4.579], Standard Error of Mean 1.553

3. Secondary Outcome: Proportion of Participants With Improvement of Fibrosis by at Least 1 Stage and/or Resolution of NASH Without Worsening of Either as Determined by Liver Biopsy
Description: Description of endpoint is Proportion of participants with improvement of fibrosis by at least 1 stage and/or resolution of NASH without worsening of either as determined by liver biopsy.
Time Frame: Week 72
Population: Due to study termination, the biopsy at Week 72 was not performed for any participants. Hence, there were no results to report.
Arm/Group | EDP-305 1.5 mg | EDP-305 2 mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Proportion of Participants With no Worsening of Fibrosis Combined With no Worsening of NASH as Determined by Liver Biopsy
Description: Proportion of participants with no worsening of fibrosis combined with no worsening of NASH as determined by liver biopsy.
Time Frame: Week 72
Population: as for outcome 1
Arm/Group | EDP-305 1.5 mg | EDP-305 2 mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Proportion of Participants With Resolution of Fibrosis as Determined by Liver Biopsy
Description: Proportion of participants with resolution of fibrosis as determined by liver biopsy at Week 72.
Time Frame: Week 72
Population: as for outcome 1
Arm/Group | EDP-305 1.5 mg | EDP-305 2 mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Proportion of Participants With Improvement in Each Histologic Feature of NASH by at Least 1 Point as Determined by Liver Biopsy
Description: Proportion of participants with improvement in each histologic feature of NASH by at least 1 point as determined by liver biopsy at Week 72.
Time Frame: Week 72
Population: as for outcome 1
Arm/Group | EDP-305 1.5 mg | EDP-305 2 mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Proportion of Participants With Improvement of Fibrosis by ≥ 2 Stages by Liver Biopsy
Description: Proportion of participants with improvement of fibrosis by ≥ 2 stages by liver biopsy.
Time Frame: Week 72
Population: as for outcome 1
Arm/Group | EDP-305 1.5 mg | EDP-305 2 mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: Proportion of Participants With Improvement in NAS by at Least 2 Points With no Worsening of Fibrosis as Determined by Liver Biopsy
Description: Proportion of participants with improvement in NAS by at least 2 points with no worsening of fibrosis as determined by liver biopsy at Week 72.
Time Frame: Week 72
Population: as for outcome 1
Arm/Group | EDP-305 1.5 mg | EDP-305 2 mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: Proportion of Participants With Improvement of Fibrosis and Resolution of NASH as a Composite Endpoint as Defined by Both Endpoints Being Met in the Same Participant
Description: Proportion of participants with improvement of fibrosis and resolution of NASH as a composite endpoint as defined by both endpoints being met in the same participant at week 72.
Time Frame: Baseline, Week 72
Population: as for outcome 1
Arm/Group | EDP-305 1.5 mg | EDP-305 2 mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0

10. Secondary Outcome: Proportion of Participants With Resolution of NASH and no Worsening of Liver Fibrosis
Description: Proportion of participants with resolution of NASH and no worsening of liver fibrosis at Week 72.
Time Frame: Week 72
Population: as for outcome 1
Arm/Group | EDP-305 1.5 mg | EDP-305 2 mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0

11. Secondary Outcome: Proportion of Participants With Histological Progression to Cirrhosis as Determined by Liver Biopsy
Description: Proportion of participants with histological progression to cirrhosis as determined by liver biopsy at Week 72.
Time Frame: Week 72
Population: as for outcome 1
Arm/Group | EDP-305 1.5 mg | EDP-305 2 mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0

12. Secondary Outcome: Participants With TEAEs Leading to Discontinuation
Description: Treatment emergent adverse events (TEAEs) were defined as AEs occurring or worsening on or after the first dose of study drug until the last dose of study drug. TEAEs were regarded as leading to discontinuation if they led to discontinuation of the study drug.
Time Frame: Day 1 to Week 72
Population: Safety population (SAF) defined as all participants who received at least one dose of study drug. Participants were included in the treatment group that corresponded to the study drug received during the study.
Measure: Count of Participants; unit: Participants
Arm/Group | EDP-305 1.5 mg | EDP-305 2 mg | Placebo
Number analyzed (Participants) | 32 | 33 | 32
Participants | 8 | 14 | 4

13. Secondary Outcome: Percentage Change of Fat in the Liver From Baseline
Description: Percentage change of fat in the liver as assessed by magnetic resonance imaging proton density fat fraction (MRI PDFF) from Baseline to Week 12.
Time Frame: Baseline, Week 12
Population: Intent-to-treat (ITT) Population:
  The ITT participants were analyzed according to the treatment to which they were randomized. The overall numbers of participants by group were N = 32, N = 33, and N = 32. The numbers of participants with available data for the specified time frame were n = 24, n =17 and n= 26 for EDP-305 1.5, 2mg and Placebo groups respectively, presented as LS Mean (95% CI).
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage change
Arm/Group | EDP-305 1.5 mg | EDP-305 2 mg | Placebo
Number analyzed (Participants) | 24 | 17 | 26
Percentage change | -25.612 [-39.387 to -11.837] | -26.069 [-40.190 to -11.948] | -14.351 [-26.908 to -1.794]
Statistical Analysis 1: Comparison: EDP-305 2 mg vs Placebo; Test type: Other; p = 0.114, ANCOVA; LS mean difference = -11.718, 95% CI 2-sided [-26.342 to 2.906], Standard Error of Mean 7.052
Statistical Analysis 2: Comparison: EDP-305 1.5 mg vs Placebo; Test type: Other; p = 0.099, ANCOVA; LS mean difference = -11.261, 95% CI 2-sided [-24.723 to 2.200], Standard Error of Mean 6.879

14. Secondary Outcome: Change in Liver Stiffness From Baseline
Description: Change in liver stiffness by magnetic resonance elastography (MRE) in kilopascal (kPa) from Baseline at Week 12.
Time Frame: Baseline, Week 12
Population: Intent-to-treat (ITT) Population:
  ITT participants were those randomized to treatment. The ITT participants were analyzed according to the treatment to which they were randomized.
  The overall numbers of participants by group were N = 32, N = 33, and N = 32. The numbers of participants with available data for the specified time frame were n = 24, n = 17 and n = 26 for EDP-305 1.5, 2mg groups and Placebo, respectively, presented as LS Mean (95% CI).
Measure: Least Squares Mean (95% Confidence Interval); unit: Kilopascal (kPa)
Arm/Group | EDP-305 1.5 mg | EDP-305 2 mg | Placebo
Number analyzed (Participants) | 24 | 17 | 26
Kilopascal (kPa) | 0.163 [-0.469 to 0.794] | 0.623 [-0.040 to 1.285] | -0.428 [-1.013 to 0.157]
Statistical Analysis 1: Comparison: EDP-305 2 mg vs Placebo; Test type: Other; p = 0.003, ANCOVA; LS mean difference = 1.050, 95% CI 2-sided [0.365 to 1.736], Standard Error of Mean 0.331
Statistical Analysis 2: Comparison: EDP-305 1.5 mg vs Placebo; Test type: Other; p = 0.064, ANCOVA; LS mean difference = 0.591, 95% CI 2-sided [-0.035 to 1.216], Standard Error of Mean 0.315

15. Secondary Outcome: Change in Triglycerides From Baseline
Description: Change in Triglycerides from Baseline at Week 12.
Time Frame: Baseline, Week 12
Population: Intent-to-treat (ITT) Population: ITT participants were those randomized to treatment. The ITT participants were analyzed according to the treatment to which they were randomized. The overall numbers of participants by group were N = 32, N = 33, and N = 32. The numbers of participants with available data for the specified time frame were n = 28, n = 26 and n=30 for EDP-305 1.5, 2mg groups and Placebo respectively.
Measure: Mean (Standard Deviation); unit: Millimoles per liter (mmol/L)
Arm/Group | EDP-305 1.5 mg | EDP-305 2 mg | Placebo
Number analyzed (Participants) | 28 | 26 | 30
Millimoles per liter (mmol/L) | -0.16 (0.725) | -0.14 (0.839) | -0.06 (0.752)

16. Secondary Outcome: Change in Adiponectin From Baseline
Description: Change in adiponectin from Baseline at Week 12.
Time Frame: Baseline, Week 12
Population: Safety population: Safety population (SAF) defined as all participants who received at least one dose of study drug. Participants were included in the treatment group that corresponded to the study drug received during the study. The overall numbers of participants by group were N = 32, N = 33, and N = 32. The numbers of participants with available data for the specified time frame were n = 27, n = 24, and n = 27 for EDP-305 1.5 mg and 2 mg groups and Placebo respectively.
Measure: Mean (Standard Deviation); unit: Micrograms per liter (µg/L)
Arm/Group | EDP-305 1.5 mg | EDP-305 2 mg | Placebo
Number analyzed (Participants) | 27 | 24 | 27
Micrograms per liter (µg/L) | 330.25 (1309.414) | -85.44 (1199.182) | 228.27 (866.829)

17. Secondary Outcome: Plasma Concentration of EDP-305
Description: Plasma concentration at second post dose (2-4 hours post dose) at Week 12.
Time Frame: 2-4 hours post dose at Week 12
Population: Pharmacokinetic (PK) Population:
  All participants receiving active study drug and having any measurable plasma concentration of study drug at any timepoint. The overall numbers of participants by group were N = 32, N = 33, and N = 32. The numbers of participants with available data for the specified time frame were n = 6 and n = 7 for EDP-305 1.5 and 2mg groups respectively.
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter (ng/mL)
Arm/Group | EDP-305 1.5 mg | EDP-305 2 mg
Number analyzed (Participants) | 6 | 7
Nanograms per milliliter (ng/mL) | 17.3783 (15.13460) | 30.0286 (24.07237)

18. Secondary Outcome: Change in VAS (Visual Analog Score) From Baseline
Description: Change in VAS from Baseline at Week 12. Change from baseline was analyzed using a restricted maximum likelihood-based MMRM technique. Two separate scales were used to assess pruritus. An itch VAS was used to record the intensity of the pruritus by Furue (Furue et al., 2013). Scale referred to no pruritus (0 point) and the end of the scale to the most severe pruritus (10 points).
  If the VAS score was greater than zero (i.e. itch), a multidimensional 5D-itch scale developed by Elman (Elman et al., 2010) indicated sum of 0-2 = score of 1, sum of 3-5 = score of 2, sum of 6-10 = score of 3, sum of 11-13 = score of 4, and sum of 14-16 = score of 5. It was used to assess five different dimensions of pruritus within the last two weeks. The five dimensions assessed were duration, degree, direction, disability, and distribution. The total 5D itch score was obtained by summing up the five domain scores and ranges between 5 (no pruritus) and 25 (most severe pruritus).
Time Frame: Baseline, Week 12
Population: Intent-to-treat (ITT) Population:
  ITT participants were those randomized to treatment. The ITT participants were analyzed according to the treatment to which they were randomized.
  The overall numbers of participants by group were N = 32, N = 33, and N = 32. The numbers of participants with available data for the specified time frame were n = 28, n = 25 and n= 30 for EDP-305 1.5, 2mg groups and Placebo, respectively, presented as LS Mean (95% CI).
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | EDP-305 1.5 mg | EDP-305 2 mg | Placebo
Number analyzed (Participants) | 28 | 25 | 30
score on a scale | 12.773 [1.386 to 24.161] | 18.548 [7.661 to 29.435] | 5.563 [-5.274 to 16.399]
Statistical Analysis 1: Comparison: EDP-305 2 mg vs Placebo; Test type: Other; p = 0.040, Mixed model repeated measures; LS mean difference = 12.986, 95% CI 2-sided [0.608 to 25.363], Standard Error of Mean 5.472
Statistical Analysis 2: Comparison: EDP-305 1.5 mg vs Placebo; Test type: Other; p = 0.242, Mixed model repeated measures; LS mean difference = 7.211, 95% CI 2-sided [-4.997 to 19.418], Standard Error of Mean 5.724

19. Secondary Outcome: Change in Total Cholesterol From Baseline
Description: Change in Total Cholesterol from Baseline to Week 12 versus placebo.
Time Frame: Baseline, Week 12
Population: Intent-to-treat (ITT) Population:
  ITT participants were those randomized to treatment. The ITT participants were analyzed according to the treatment to which they were randomized. The overall numbers of participants by group were N = 32, N = 33, and N = 32. The numbers of participants with available data for the specified time frame were n = 28, n = 26, and n = 30 for EDP-305 1.5, 2 mg groups and Placebo respectively.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | EDP-305 1.5 mg | EDP-305 2 mg | Placebo
Number analyzed (Participants) | 28 | 26 | 30
mmol/L | 0.07 (0.977) | -0.07 (1.116) | 0.00 (0.946)

20. Secondary Outcome: Change in HDL From Baseline
Description: Change in HDL from Baseline at week 12.
Time Frame: Baseline, Week 12
Population: Intent-to-treat (ITT) Population:
  ITT participants were those randomized to treatment. The ITT participants were analyzed according to the treatment to which they were randomized. The overall numbers of participants by group were N = 32, N = 33, and N = 32. The numbers of participants with available data for the specified time frame were n = 27, n = 25, and n = 30 for EDP-305 1.5, 2 mg groups and Placebo respectively.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | EDP-305 1.5 mg | EDP-305 2 mg | Placebo
Number analyzed (Participants) | 27 | 25 | 30
mmol/L | -0.08 (0.200) | -0.11 (0.255) | 0.01 (0.149)

21. Secondary Outcome: Change in LDL From Baseline
Description: Change in LDL From Baseline to Week 12.
Time Frame: Baseline, Week 12
Population: Intent-to-treat (ITT) Population:
  ITT participants were those randomized to treatment. The ITT participants were analyzed according to the treatment to which they were randomized. The overall numbers of participants by group were N = 32, N = 33, and N = 32. The numbers of participants with available data for the specified time frame were n = 28, n = 26, and n = 30 for EDP-305 1.5 mg, 2mg groups and Placebo respectively.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | EDP-305 1.5 mg | EDP-305 2 mg | Placebo
Number analyzed (Participants) | 28 | 26 | 30
mmol/L | 0.24 (0.856) | 0.08 (0.949) | -0.03 (0.835)

ADVERSE EVENTS:
Time Frame: Day 1 to Week 72
Description: Treatment emergent adverse events were defined as AEs occurring or worsening on or after the first dose of study drug until the last dose of study drug.
Arm/Group | EDP-305 1.5 mg | EDP-305 2 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/33 | 0/32
Serious Adverse Events (participants affected / at risk) | 2/32 | 0/33 | 0/32
Other Adverse Events (participants affected / at risk) | 28/32 | 31/33 | 20/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | EDP-305 1.5 mg (N=32) | EDP-305 2 mg (N=33) | Placebo (N=32)
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | EDP-305 1.5 mg (N=32) | EDP-305 2 mg (N=33) | Placebo (N=32)
Pruritus (Skin and subcutaneous tissue disorders) | 25 | 25 | 12
Rash (Skin and subcutaneous tissue disorders) | 3 | 2 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Blood creatine phosphokinase increased (Investigations) | 2 | 1 | 0
Lipase increased (Investigations) | 0 | 2 | 2
Abdominal pain upper (Gastrointestinal disorders) | 2 | 4 | 1
Nausea (Gastrointestinal disorders) | 2 | 1 | 3
Toothache (Gastrointestinal disorders) | 0 | 0 | 2
Headache (Nervous system disorders) | 2 | 3 | 2
Dizziness (Nervous system disorders) | 2 | 3 | 1
Fatigue (General disorders) | 2 | 3 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 3
Abdominal pain (Gastrointestinal disorders) | 3 | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1 | 2
Abdominal pain lower (Gastrointestinal disorders) | 2 | 1 | 0
Urinary tract infection (Infections and infestations) | 4 | 3 | 4
COVID-19 (Infections and infestations) | 3 | 1 | 1
Blood pressure increased (Investigations) | 0 | 0 | 2
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2
Post vaccination syndrome (Injury, poisoning and procedural complications) | 0 | 0 | 2
Hypertension (Vascular disorders) | 1 | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2

LIMITATIONS AND CAVEATS:
No limitations reported for the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2021-03-21): https://cdn.clinicaltrials.gov/large-docs/10/NCT04378010/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-14): https://cdn.clinicaltrials.gov/large-docs/10/NCT04378010/SAP_001.pdf